CLINICAL TRIAL: NCT01631292
Title: A Pilot Dose Response Study to Vitamin D in Obesity and Weight Loss: Effect on Bone
Brief Title: Vitamin D Supplementation in Obesity and Weight Loss (3DD Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers University (Other)
Responsible Party: Principal Investigator, Sue A. Shapses, Ph.D., RD, Professor, Rutgers University
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: BBGP201095157
Record Dates: First submitted 2011-06-30; First posted 2012-06-29 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 600 IU D3 (Placebo Comparator)
  Interventions: Dietary Supplement: 600 IU Vitamin D3
- 2000 IU D3 (Active Comparator)
  Interventions: Dietary Supplement: 2000 IU Vitamin D3
- 4000 IU D3 (Active Comparator)
  Interventions: Dietary Supplement: 4000 IU Vitamin D3

INTERVENTIONS:
Dietary Supplement: 600 IU Vitamin D3 — Once daily
  Arms: 600 IU D3
Dietary Supplement: 2000 IU Vitamin D3 — Once daily
  Arms: 2000 IU D3
Dietary Supplement: 4000 IU Vitamin D3 — Once daily
  Arms: 4000 IU D3

SUMMARY:
In this study, we will provide supplemental vitamin D in postmenopausal overweight/obese women, and hypothesize that it will not affect areal BMD, but will alter bone compartments (trabecular and cortical bone). In addition, higher vitamin D intake will increase serum 25OHD and suppress serum PTH and bone turnover during weight reduction. Secondary outcomes include the influence of vitamin D and weight loss on markers of insulin resistance and on cognitive tests of attention, learning, and memory.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index of 25-40 kg/m2
* Postmenopausal
* Age 50-72 years

Exclusion Criteria:

* Women who are taking any medication known to influence Calcium or bone metabolism,
* Evidence of diseases known to influence Calcium metabolism (i.e. metabolic bone disease)
* hyperparathyroidism
* untreated thyroid disease
* significant immune disease
* hepatic disease
* renal disease or a kidney stone in the last 5 years
* significant cardiac disease
* active malignancy or cancer therapy within the past year

Ages: 50 Years to 72 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2010-01; Primary Completion 2015-05 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Bone mineral density (BMD) | 1 year
  BMD
Bone quality | 1 year
  thickness (mm)

SECONDARY OUTCOMES:
Bone turnover markers | Baseline, 6 months, 12 months
  osteocalcin (others include PINP and CTX)
Glycemic indices | Baseline, 6 months and 12 months
  glucose and insulin
Cognition and biochemical markers | One year
  Cognitive measures and serum biochemical markers
cholesterol absorption | baseline and one year
  Serum levels
serum vitamin D | Baseline, 6 months and 12 months
  25(OH)D
Bone regulating hormones | Baseline, 6 months and 12 months
  PTH

CONTACTS AND LOCATIONS:
Overall Officials: Sue Shapses, PhD, Principal Investigator — Rutgers University
Locations (1):
- Rutgers University- Thompson Hall, New Brunswick, New Jersey, United States

REFERENCES:
- [Background] Castle M, Fiedler N, Pop LC, Schneider SJ, Schlussel Y, Sukumar D, Hao L, Shapses SA. Three Doses of Vitamin D and Cognitive Outcomes in Older Women: A Double-Blind Randomized Controlled Trial. J Gerontol A Biol Sci Med Sci. 2020 Apr 17;75(5):835-842. doi: 10.1093/gerona/glz041. PMID 30951148
- [Background] Pop LC, Sukumar D, Schneider SH, Schlussel Y, Stahl T, Gordon C, Wang X, Papathomas TV, Shapses SA. Three doses of vitamin D, bone mineral density, and geometry in older women during modest weight control in a 1-year randomized controlled trial. Osteoporos Int. 2017 Jan;28(1):377-388. doi: 10.1007/s00198-016-3735-z. Epub 2016 Aug 17. PMID 27535752
- [Derived] Ogilvie AR, Schlussel Y, Sukumar D, Meng L, Shapses SA. Higher protein intake during caloric restriction improves diet quality and attenuates loss of lean body mass. Obesity (Silver Spring). 2022 Jul;30(7):1411-1419. doi: 10.1002/oby.23428. Epub 2022 May 11. PMID 35538903